CLINICAL TRIAL: NCT06388746
Title: Minimal Intervention Techniques for Arresting Caries in Primary Molars: a Randomized Clinical Trial With 12 Months Follow-up.
Brief Title: Arresting Carious Lesions With Minimal Intervention Techniques
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Sotiria Gizani, Associate Professor, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NKUA
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Caries,Dental
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caries removal group (Experimental): Cavitated lesion will be isolated with cotton rolls and air-dried. Gel will be placed in the cavity and kept there for 60 seconds to allow for the decayed tissue to become softer. The softened tissue will be removed with a hand instrument. The gel will be reapplied, until complete removal of the carious tissue is achieved. Teeth will be restored using a high viscosity glass ionomer cement.
  Interventions: Other: BRIX3000®
- Caries arrest group (Active Comparator): Cavitated lesion will be isolated with cotton rolls and air-dried. One drop of component 1 (38% Silver Fluoride (AgF) in water) will be applied for 60 seconds using a microbrush, followed by two drops of component 2 (potassium iodide) for 90 seconds. Teeth will be restored using a high viscosity glass ionomer cement.
  Interventions: Other: Riva Star Aqua, SDI Limited, Australia

INTERVENTIONS:
Other: BRIX3000® — A gel that when applied to the tooth completely removes carious tissues in a chemo mechanical way without rotary instruments. It contains an enzyme that has bactericidal, bacteriostatic and anti-inflammatory properties and proteolytic properties that help soften and break down decayed tissue without destroying the underlying healthy collagen fibers.
  Arms: Caries removal group
Other: Riva Star Aqua, SDI Limited, Australia — A solution that contains 44,800 ppm F and 253,870 ppm Ag. It acts as a fluoride storage for the acid challenges, while inhibites demineralization of hydroxyapatite crystals and preserves collagen from degradation in demineralized tissues.
  Arms: Caries arrest group

SUMMARY:
A single-blinded randomized clinical trial with a split-mouth design that will assess the 12-month clinical and radiographic success of two minimally invasive treatment techniques, one using a chemo-mechanical caries removal agent and one using a caries arresting agent, for the treatment of deep caries in primary molars.

DETAILED DESCRIPTION:
Fifty children (100 teeth) aged 4 to 8 years with a non-contributary medical history and at least two carious primary molars (ICDAS 5 and 6) on different quadrants will be randomly assigned to either treatment group, using computer-generated numbers.

Each cavitated lesion will be isolated with cotton rolls and air-dried before being treated with one of the two types of minimal intervention technique according to the manufacturer's instructions. After the application of the agents all teeth will be restored using a high viscosity glass ionomer cement.

Patients will be followed clinically at 6 and 12 months and radiographically at 12 months to evaluate success of the procedures.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4 to 8 years with a non-contributary medical history and sufficient compliance for the caries treatment will be included. The eligible children should have at least two carious primary molars (cavitated lesions up to 2/3 of dentin, corresponding to ICDAS 5 and 6) on different quadrants without any periapical pathology detected radiographically.

Exclusion Criteria:

* Children aged below 4 years and above 8 years, with compromised medical history and/or allergies, with clinical or radiographic signs or symptoms of pulp pathology and with developmental dental defects will be excluded.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
clinical success | 6 and 12 month post-treatment
  Presence/absence of: tooth pain, swelling, abscess, fistula, mobility, tenderness to percussion, tenderness to palpation.
radiographic success | 12 month post-treatment
  Presence/absence of: periapical pathology, pulp canal obliteration, root resorption, secondary caries formation.

SECONDARY OUTCOMES:
Longevity and the quality of the final restoration | 6 and 12 months post-treatment
  Evaluation of retention, marginal integrity, marginal discoloration, anatomic form and secondary caries using USPHS criteria.
Patient's acceptance | immediately post-treatment
  intensity or frequency of various symptoms, such as pain using the Visual Analogue Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Sotiria Gizani, Assoc Prof, Principal Investigator — Department Of Paediatric Dentistry, National And Kapodistrian University Of Athens